CLINICAL TRIAL: NCT03010475
Title: A Trial Investigating the Effect of Oral Semaglutide on the Pharmacokinetics of Furosemide and Rosuvastatin in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4250; 2015-003908-23 (EudraCT Number); U1111-1173-8618 (Other: UTN)
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Furosemide; Rosuvastatin Calcium; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furosemide/Rosuvastatin/SNAC/Semaglutide (Experimental)
  Interventions: Drug: Furosemide; Drug: Rosuvastatin; Drug: SNAC; Drug: Semaglutide

INTERVENTIONS:
Drug: Furosemide — Oral administration A total of three single doses.
Drug: Rosuvastatin — Oral administration. A total of three single doses.
Drug: SNAC — Oral administration. A total of five single doses.
Drug: Semaglutide — Oral administration. Once daily.

SUMMARY:
This trial is conducted in Europe. Tha aim of this trial is to investigate the effect of oral semaglutide on the pharmacokinetics of furosemide and rosuvastatin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 20.0-29.9 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiography and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Smoker (defined as a subject who is smoking at least one cigarette or the equivalent per day)
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Have personal or family history of myopathy
* Previous history of muscular toxicity with another HMG-CoA reductase inhibitor or fibrate
* Thyroid-Stimulating Hormone outside lower limit of normal minus 10 percent and upper limit of normal plus 10 percent
* Creatine kinase above 5 x upper limit of normal
* Asian subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Area under the furosemide plasma concentration-time curve | day 1, day 7, day 54
  Based on sampling between 0 and 12 hours
Area under the rosuvastatin plasma concentration-time curve | day 2, day 8, day 55
  Based on sampling between 0 and 96 hours

SECONDARY OUTCOMES:
Maximum observed furosemide plasma concentration | day 1, day 7, day 54
Maximum observed rosuvastatin plasma concentration | day 2, day 8, day 55

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Jordy AB, Albayaty M, Breitschaft A, Anderson TW, Christiansen E, Houshmand-Oregaard A, Manigandan E, Baekdal TA. Effect of Oral Semaglutide on the Pharmacokinetics of Levonorgestrel and Ethinylestradiol in Healthy Postmenopausal Women and Furosemide and Rosuvastatin in Healthy Subjects. Clin Pharmacokinet. 2021 Sep;60(9):1171-1185. doi: 10.1007/s40262-020-00976-x. PMID 33782832